CLINICAL TRIAL: NCT04403477
Title: Convalescent Plasma Transfusion Therapy in Severe COVID-19 Patients- a Tolerability, Efficacy and Dose-response Phase II RCT
Brief Title: Convalescent Plasma Therapy in Severe COVID-19 Infection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Collaborators: Dhaka Medical College (Other)
Responsible Party: Principal Investigator, Fazle Rabbi Chowdhury, Assistant Professor, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BSMMU/2020/6104
Record Dates: First submitted 2020-05-20; First posted 2020-05-27 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Covid19; Convalescence
MeSH Terms: conditions — COVID-19; Convalescence | interventions — Immunization, Passive

STUDY DESIGN:
Intervention Model Description: Arm-A: Standard supportive treatment; Arm-B: Standard supportive treatment + CP 200 ml; Arm C: Standard supportive treatment + CP 400 ml
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard treatment (No Intervention): Standard supportive treatment (Oxygen, Enoxaparine, antibiotic, fluid, immune modulator (Steroid) and or antiviral (favipiravir or ramdesivir or lopinavir + ritonavir)
- Standard treatment + 200 ml plasma (Experimental): Standard supportive treatment + 200 ml apheretic convalescent plasma single transfusion
  Interventions: Biological: Convalescent plasma
- Standard treatment + 400 ml plasma (Experimental): Standard supportive treatment + 400 ml apheretic convalescent plasma single transfusion
  Interventions: Biological: Convalescent plasma

INTERVENTIONS:
Biological: Convalescent plasma — Apheretic convalescent plasma from a COVID-19 survivor
  Other Names: Plasma therapy
  Arms: Standard treatment + 200 ml plasma; Standard treatment + 400 ml plasma

SUMMARY:
As of March 18, 2020, COVID-19 cases were reported in approximately 195 countries. No specific therapeutic agents or vaccines for COVID-19 are available. Several therapies, such as remdesivir and favipiravir, are under investigation, but the antiviral efficacy of these drugs is not yet known. The use of convalescent plasma (CP) was recommended as an empirical treatment during outbreaks of Ebola virus in 2014. A protocol for treatment of Middle East respiratory syndrome coronavirus (MERS-CoV) with CP was established in 2015. This approach with other viral infections such as SARS-CoV, H5N1 avian influenza, and H1N1 influenza also suggested that transfusion of CP was effective. In previous reports, most of the patients received the CP by single transfusion. In a study involving patients with pandemic influenza A(H1N1) 2009 virus infection, treatment of severe infection with CP (n = 20 patients) was associated with reduced respiratory tract viral load, serum cytokine response, and mortality. In another study involving 80 patients with SARS, the administration of CP was associated with a higher rate of hospital discharge at day 22 from symptom onset compared with patients who did not receive CP. Accordingly, these findings raise the hypothesis that use of CP transfusion could be beneficial in patients infected with SARS-CoV-2. The objective of this study is to describe the initial clinical experience with CP transfusion administered to severe COVID-19 patients. The primary endpoint of this trial would be to assess the tolerability, efficacy, and dose-response of CP in severe COVID-19 patients. The secondary endpoint would be to assess the clinical and laboratory parameters after therapy, in-hospital mortality, length of hospital stay, reduction in the proportion of deaths, length of ICU stay, requirement of ventilator and duration of ventilator support. All RT-PCR positive cases with features of severe infection will be enrolled in this study. Apheretic CP will be collected from a recovered patient (consecutive two RT-PCR samples negative) between day 22 to 35 days of recovery and those with the antibody titre above 1:320.

This RCT will consist of three arms, a. standard care, b. standard care and 200 ml CP and c. standard care and 400 ml CP as a single transfusion. Twenty (20) patients will be enrolled for each arm. Randomization will be done by someone not associated with the care or assessment of the patients by means of a random number table. Allocations will be concealed in sequentially numbered, opaque, sealed envelopes. Clinical parameters [fever, cough, dyspnea, respiratory rate, PaO2/ FiO2 level, pulse, BP, the requirement of O2, and others] will be recorded before and after CP. Laboratory parameters such as complete blood count, CRP, chest X-ray, SGPT, SGOT, S. Ferritin, and serum antibody titre will be measured before and after transfusion. Allergic or serum sickness-like reactions will be noted and adjusted with outcome. Laboratory tests including RT-PCR will be done at BSMMU virology and laboratory medicine department. Apheretic plasma will be collected at the transfusion medicine department of SHNIBPS hospital, ELISA, antibody titre will be done at CMBT, and patients will be enrolled at DMC and MuMCH. All necessary screening tests will be done before transfusion.

Graphpad Prism v 7.0 will be used for analysis. One way ANOVA test, a non-parametric Mann-Whitney test, and a Kruskal-Wallis test will be performed to compare the arms. For parametric outcomes, the investigators will compare the odds ratios across the pairs.

DETAILED DESCRIPTION:
Rationale of the Study Currently no specific treatment is available against COVID-19 infection. Supportive treatment along with concentrated oxygen is the only mean of treatment. Researchers have already opened over 180 clinical trials of potential COVID-19 treatments for recruitment, and nearly 150 could start soon. However, to date, no clinical intervention trial has been completed and reported. Based on anecdotes (small case series), some of the promising drugs could be azithromycin - hydroxychloroquine combination, Lopinavir/ Ritonavir, Tocilizumab, Ramdisivir, Favirinapir, and others. CP transfusion is another promising option, which had been tried before in SARS-CoV, MERS-CoV, and Flu and Ebola viral infection. Its effectiveness against COVID-19 yet not explored. A recently published case series consists of ten cases that forecast promising results. Therefore, a phase II RCT to explore the tolerability, efficacy, and dose-response needs to explore urgently.

The cases started to escalate in Bangladesh and the number of confirmed cases already crossed a thousand marks. Considering the cost and shortage of other above mentioned anti-viral and biologics, it is inevitable that many of our patients possibly could not afford or get it. However, the CP can be easily collected from the recovered patients and can easily be processed to use it against active infection. This could be an effective and cheap treatment option for a country like ours to face this catastrophe. Therefore conducting a phase II RCT on CP transfusion is the demand of time.

Research question:

Does CP transfusion is tolerable and effective in treating severe COVID-19 patients compared to standard treatment?

Objectives:

General Objective:

To assess the tolerability, efficacy, and dose-response of CP transfusion in severe COVID-19 patients

Specific Objectives:

1. To identify the appropriate effective dose of CP therapy
2. To identify the efficacy of the therapy with their endpoint
3. To examine the clinical improvement after CP transfusion in severe COVID-19 patients
4. To assess the laboratory improvement after CP transfusion in severe COVID-19 patients

Study design:

Phase II RCT

Place of study:

Bangabandhu Sheikh Mujib Medical University (BSMMU), Sheikh Hasina Burn & Plastic Surgery Institute, Dhaka Medical College, Mugda Medical College and Centre for Medical Biotechnology

Study period:

May 2020 - October 2020 (Six months)

Study population:

COVID=19 positive patients who are diagnosed on the basis of RT-PCR at BSMMU fever clinic or by any other government-designated laboratory and admitted at DMCH, MuMC, and BSMMU.

Randomization and blinding method:

Randomization will be done by someone not associated with the care or assessment of the patients by means of a random number table. Allocations will be concealed in sequentially numbered, opaque, sealed envelopes. In this pilot study, the CP or standard care will not be blinded. However, the primary outcome (oxygen saturations, PaO2/FiO2, and BP) will be recorded using an objective automated method; the study staff will not be able to influence the recording of these data.

Sample size:

No similar study has been performed previously. Therefore no data are available that could be used to generate a sample size calculation. This pilot study is required to provide some initial data on efficacy and safety that will allow the design of a larger study.

Research instruments

1. General questionnaire for assessing socio-demographic data.
2. A checklist of clinical findings
3. A checklist of investigation findings.

Measures of Variables

1. Socio-Demographic variables

   * Age
   * Gender (Male/Female)
   * Living area (Urban/Rural)
   * Occupation
2. Clinical variables:

   * Symptoms
   * Systolic blood pressure (in mmHg)
   * Diastolic blood pressure (in mmHg)
   * Temperature
   * Respiratory rate
   * Heart rate
   * GCS
3. Laboratory variables

   * CXR
   * CBC
   * CRP
   * S. Ferritin
   * SGPT
   * SGOT
   * Antibody titre

Procedure of collection of Apheretic plasma

1. Pre-donation screening: First of all, 3 ml blood will be drawn from peripheral venous site preferably from dorsum of the hand, and will be kept in EDTA tube for further testing. Blood group will be confirmed by using known antisera. Screening test of 5 diseases (HBs Ag , Anti HCV, HIV, Syphilis, and Malaria) will be tested by the device method. An automated analyzer will count complete blood count. If all things remain favorable, the next step will be followed.
2. Safety assessment: Body weight and height of the donor will be measured by a conventional method (standard digital weight and height scale). For preventing citrate toxicity or hypocalcaemic complications (twitching, numbness, nausea, mild respiratory difficulty, etc) 500 mg calcium carbonate will be given to every donor before starting the procedure. Blood pressure and pulse will be monitored in every 10-minute interval for precaution throughout the procedure. Weight, height, and CBC parameter will be given in apheresis machine for setting up. Visible and easily palpable anti cubital vein will be selected for venepuncture. Before puncturing the vein, at least 50-60 mm of Hg pressure will be given above the venepuncture area for maintaining sustained pressure. When everything is ready, the procedure will be started by puncturing a single needle in a targeted vein.

Steps of Convalescent Plasma (CP) transfusion Before giving CP to the patient blood pressure, pulse, temperature, the respiratory rate will be recorded. It can be given through the central venous catheter or by peripheral channel. If peripheral venous site chosen then at least 21g needle should be confirmed. Blood group and cross-matching should be confirmed before starting the transfusion. When there is no chance of clerical mistake then CP transfusion can be started at the rate of 100 ml/hour.

Safety Assessment:

If patient was suffering from fever then a temperature chart should be maintained. When the temperature will be raised above 2 degrees Fahrenheit from the baseline then transfusion should be stopped and antipyretic should be given according to the body weight. After a pause of 10 minutes, transfusion can be started. If patient, feels excessive itching specific area or whole over the body then Injection Chlorpheniramine maleate will be given. The steroid would be preserved for managing severe respiratory distress or uncontrollable itching. Blood pressure, pulse, and respiratory will be monitored every 30 minutes interval regularly.

The procedure of measuring antibody titre

SARS-CoV-2 IgG antibody titer will be tested by ELISA according to the following protocol:

1. At first the serum/plasma samples (10μL) were diluted to 1:40, 1:80, 1:160, 1:320, and 1:640 by serial dilution.
2. 100μl of sample diluents will be added into each well (except blank and control well) which are pre-coated with SARS-CoV-2 antigens.
3. Then 10μl of specimen will be added. 100μl controls will be added to the assigned well directly. All samples will be run in duplicate.
4. The plate will be covered with the plate cover and will be incubated for 30 minutes at 37°C.
5. At the end of the incubation, each well will be washed 5 times with diluted Wash Buffer.
6. 100μl of conjugate will be added into each well except the Blank.
7. Incubation for 20 minutes at 37°C.
8. At the end of the incubation, each well will be washed 5 times with diluted Wash Buffer.
9. 50μl of Substrate Solution A and 50μl of Substrate Solution B will be added into each well. Incubation for 10 minutes at 37°C avoiding light.
10. 50μl of Stop Solution will be added into each well.
11. The plate reader will be calibrated with the Blank well and the absorbance will be read at 450nm.
12. The sample OD value was ≥cutoff OD value will indicate IgG antibody positive.
13. The IgG antibody titre will be determined by endpoint dilution.

Due to lack of COVID-19 plasmid in Bangladesh and global shortage, 2 ml seum will be preserves from each donor and later shipped to peter Medawar building for pathogen research, University of Oxford. Research collaborators in Oxford will conduct the neutralizing antibody titre and the investigators will later match them with each donor. The expenses for neutralizing antibody titre test will be managed by the Oxford colleagues.

Statistical analysis:

Graphpad Prism v 7.0 will be used for analysis. Demographic factors and clinical characteristics will be summarized with counts (%) for categorical variables and median (interquartile range [IQR]) for continuous variables, as none was expected to be normally distributed. The main analysis will be carried out on an intention-to-treat basis. For the primary outcome, the investigators will compare the mean between three arms using a one-way ANOVA test. The investigators will also do posthoc analysis in Prism assessing (log-rank Mantel-Cox test) time to sustained saturations >93% and PaO2/FiO2<200 mm of Hg censored during enrolment, 3 days and 7 days after enrolment in a single time point. For non-parametric secondary outcomes, all groups will be compared using a Kruskal-Wallis test; if significant, the investigators then planned to perform pairwise comparisons with a non-parametric Mann-Whitney test. For parametric outcomes, the investigators compared the odds ratios across the pairs.

Facilities and procedure:

The RT-PCR and other study-related testing will be done at BSMMU. BSMMU fever clinic already treated more than 1200 COVID-19 positive cases. Potential donors will be tracked from this patient pool. Donors who will agree and give consent will be then sent to the Transfusion medicine department of SHBPSI. 5 ml plasma will be collected and sent to the CMBT laboratory for ELISA based antibody titre. If the titre fulfills the desired level (1:320 and above), then 200 ml or 400 ml apheretic plasma (depending on availability and consent of the donor) will be collected on the next day. 5 ml serum will be also be collected for sending into the Peter Medawar Building for Pathogen Research, Oxford University for checking the neutralizing antibody titre. This will be sent later and matched with the donor. The samples will be shipped under the coverage of the materials transfer agreement (MTA). Dr. Fazle Rabbi Chowdhury, the Co-PI of this project have the necessary permission for shipping samples overseas. In the final stage, the CP will be handover to the clinical team at DMCH and MuMCH as per their demand for transfusion. The clinical team will ensure the laboratory sample collection before and after CP transfusion and will record the data in the case record form. A laboratory medicine team of BSMMU will support the clinical team for lab testing.

ELIGIBILITY:
Inclusion Criteria:

1. Respiratory rate > 30 breaths/min; PLUS
2. Severe respiratory distress; or SpO2 ≤ 88% on room air or PaO2/FiO2≤ 300 mm of Hg, PLUS
3. Radiological evidence of bilateral lung infiltrate, AND OR
4. Systolic BP < 90 mm of Hg or diastolic BP <60 mm of Hg. AND OR
5. Criteria 1 to 4 AND or patient in Ventilator support

Exclusion Criteria:

1. Patients below18 years.
2. Pregnant women and breast-feeding mothers.
3. Previous history of allergic reaction to plasma
4. Those who will not give consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-05-20 (Actual); Primary Completion 2020-07-20 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of In-hospital mortality | 7 days
  % of patients died after enrolment
Time to death | 7 days
  Time to death in hours after enrolment

SECONDARY OUTCOMES:
Fever | 7 days
  Temperature in degree Fahrenheit at Day 0, 1, 3, 7
Respiratory distress | 7 days
  Respiratory rate per minute at Day 0, 1, 3, 7
Saturation of oxygen | 7 days
  Saturation of oxygen in % at Day 0, 1, 3, 7
Blood pressure | 7 days
  Blood pressure in mm of Hg at Day 0, 1, 3, 7
Oxygen requirement | 7 days
  Oxygen requirements in liter/min at Day 0, 1, 3, 7
C-reactive Protein | Day 0, 3 and 7
  CRP level in mg/litre
Ferritin | Day 0, 3 and 7
  Serum Ferritin level in ng/ml
SGPT | Day 0, 3 and 7
  Serum SGPT level in I/U
SGOT | Day 0, 3 and 7
  Serum SGOT level in I/U
ICU stay | 14 days
  Duration of ICU stay in days
Ventilator support | 14 days
  Requirement of ventilator support in hours
Hospital stay | 14 days
  Duration of hospital stay in days
Proportion of Transfusion reaction | 24 hours
  % of patients developed early transfusion reaction like fever, sweating, rash, abdominal pain, urticaria, vomiting, wheezing, chest tightness and hypotension

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad S Rahman, MPhil; FCPS, Study Chair — Professor and Chairman of Pharmacology, BSMMU
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with the journal authority and make public as part of the publication
Supporting Information: SAP, ICF, CSR
Time Frame: six months
Access Criteria: Available on public domain like figshare, researchgate and others

REFERENCES:
- [Derived] Chowdhury FR, Hoque A, Chowdhury FUH, Amin MR, Rahim A, Rahman MM, Yasmin R, Amin MR, Miah MT, Kalam MA, Rahman MS. Convalescent plasma transfusion therapy in severe COVID-19 patients- a safety, efficacy and dose response study: A structured summary of a study protocol of a phase II randomized controlled trial. Trials. 2020 Oct 26;21(1):883. doi: 10.1186/s13063-020-04734-z. PMID 33106167